CLINICAL TRIAL: NCT01255631
Title: Use of Pulsed Electromagnetic Fields in Reducing Arm and Shoulder Complaints in Breast Cancer Patients After Lymph Node Dissection
Brief Title: Pulsed Electromagnetic Fields (PEMF) and Post-Axillary Surgery Morbidity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Christine Hsu Rohde, MD, Assistant Professor of Clinical Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAE3803
Record Dates: First submitted 2010-12-01; First posted 2010-12-07 (Estimated); Results first posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Shoulder Symptoms After Lymph Node Dissection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham PEMF device (Sham Comparator)
  Interventions: Device: Sham PEMF Device
- PEMF Device (Active Comparator)
  Interventions: Device: PEMF Device

INTERVENTIONS:
Device: PEMF Device — The PEMF device we will use in this study is FDA approved for "adjunctive use in the palliative treatment of post-operative pain and edema in superficial soft tissue" (510(k) number: K903675). There are no side effects to use of a PEMF device. In the treatment arm, the PEMF would be automatically delivered for 15 minutes every two hours for one month. The manufacturer (Ivivi Technologies, Inc., Northvale, NJ) has already designed a lightweight, disposable device that can be placed around the patient's arm and taped in place. The patient would keep the device in place for two weeks, when they return for a followup visit and receive a fresh device to wear for an additional two weeks.
  Other Names: Ivivi Sofpulse Torino
  Arms: PEMF Device
Device: Sham PEMF Device — Inactive PEMF device, delivers no PMF
  Arms: Sham PEMF device

SUMMARY:
The most important prognostic indicator for the breast cancer patient is the axillary lymph node status. With the introduction of the sentinel lymph node biopsy, many women were spared the morbidity of a full axillary lymph node dissection(ALND) while having the axillary nodes assessed with a low false negative rate. Approximately 30% of women who undergo ALND experience shoulder/arm morbidity including numbness, pain, weakness and decreased range of motion. In addition, the sentinel lymph node dissection (SLND) held the promise that women with early stage breast cancer would be able to avoid the dreaded morbidity associated with axillary lymph node dissections including lymphedema, decreased range of motion and pain. Since the adoption of SLN, numerous papers have documented that SLN is superior to ALND. However, patients who undergo SLN still have a significant amount of pain with this procedure. There are few published studies which objectively assess the subjective and objective symptoms of SLND.

Pulsed electromagnetic fields (PEMF) have been shown to be effective in the treatment of fractures and spinal fusion, relief of pain in acute sprains and whiplash injuries, improvement of skin blood flow, healing of venous stasis ulcers, and reduction of postmastectomy lymphedema. Indeed, radiofrequency PEMF devices are FDA approved for pain and edema relief. PEMF devices are economical and disposable, and can be incorporated unobtrusively in standard post-op dressings. We have recently reported, in a double-blind, placebo-controlled study on breast reduction, that post-op PEMF therapy produced a significant decrease in pain and pain medication use, along with a concomitant decrease in IL1-beta in the wound bed.1 The current pilot study will be designed to determine if PEMF treatment, given in addition to standard of care, can reduce post-operative discomfort and morbidity after lumpectomy and SLND, or lumpectomy and ALND. Lumpectomy and ALND/SLND patients enrolled in the double-blind, placebo-controlled study will undergo standard surgery, but will be randomized to one of two groups: the treatment group with a PEMF coil placed around the arm and the control group with a coil that delivers no PMF. We expect postoperative pain to be reduced in the PEMF-treated patients as well as improved arm mobility and strength. The use of PEMF might reduce the need for narcotic pain medications and their side effects of sedation, nausea, and vomiting. It may also reduce costs related to arm morbidity.

DETAILED DESCRIPTION:
In the treatment arm, the PEMF would be automatically delivered for 15 minutes every two hours for one month. The manufacturer (Ivivi Technologies, Inc., Northvale, NJ) has already designed a lightweight, disposable device that can be placed around the patient's arm and taped in place. The patient would keep the device in place for two weeks, when they return for a followup visit and receive a fresh device to wear for an additional two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include patients undergoing axillary lymph node dissection or sentinel lymph node dissection for breast cancer. Patients undergoing lumpectomy with the axillary surgery will be included.

Exclusion Criteria:

* Patients undergoing mastectomy with the axillary surgery will be excluded.
* Patients with prior axillary radiation or prior arm impairment will be excluded.
* Patients with pacemakers will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rohde, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Helms G, Kuhn T, Moser L, Remmel E, Kreienberg R. Shoulder-arm morbidity in patients with sentinel node biopsy and complete axillary dissection--data from a prospective randomised trial. Eur J Surg Oncol. 2009 Jul;35(7):696-701. doi: 10.1016/j.ejso.2008.06.013. Epub 2008 Oct 5. PMID 18838245
- [Background] Rohde C, Chiang A, Adipoju O, Casper D, Pilla AA. Effects of pulsed electromagnetic fields on interleukin-1 beta and postoperative pain: a double-blind, placebo-controlled, pilot study in breast reduction patients. Plast Reconstr Surg. 2010 Jun;125(6):1620-1629. doi: 10.1097/PRS.0b013e3181c9f6d3. PMID 20527063

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sham PEMF Device | PEMF Device
Started | 13 | 9
Completed | 4 (study terminated due to poor enrollment) | 3 (study terminated due to poor enrollment)
Not Completed | 9 | 6
Not completed — poor enrollment, no data analyzed | 9 | 6

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was determined by the patients who completed the study (7 total patients: 4 Sham and 3 active PEMF)
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham PEMF Device | PEMF Device | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Level on Visual Analog Scale
Description: Pain will be the primary outcome measured by patient level of pain as quantified by a visual analog scale with written descriptions, and amount of pain medication used hourly until the patient is discharged (up to a maximum of six hours post-op), then daily for a total of two weeks post-op. The VAS pain scale ranges from 0 (no pain) to 10 (worst possible pain).
Time Frame: 2 weeks
Population: Only 7 patients completed the study by quantifying the level of their pain post-operatively on a visual analog scale from 0-10. The medication logs and two week post-op analogs could not be utilized for the analysis since all 7 patients did not complete these logs.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 4 | 3
units on a scale | 3.878 (2.811) | 5.239 (2.979)

2. Secondary Outcome: Jackson Pratt (JP) Drain Output
Description: Total volume (in units of millimeters - mL) of Jackson Pratt (JP) drain output on post-operative day 1 and day 2 were recorded for patients in the study.
Time Frame: Post-Operative Day 1 & 2 (2 Days)
Population: For the 7 patients who completed the study, the mean and standard deviations for the total JP drain output (in milliliters - mL) from post-operative days 1 & 2 (2 days total) were analyzed as a secondary outcome.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 4 | 3
milliliters (mL) | 136.5 (74.633) | 85.333 (39.272)

3. Secondary Outcome: Patient Self-Assessment of Shoulder and Arm Symptoms Before and After PEMF
Description: No participants were assessed for this secondary outcome measure: patient self-assessment of shoulder and arm symptoms before and after PEMF. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. Patients did not complete the necessary surveys assessing their shoulder and arm symptoms; therefore, no meaningful results could be derived since there were no surveys to compare before and after PEMF data points.
Time Frame: Pre- and Post-Operative Period
Population: No participants were assessed for this secondary outcome measure: patient self-assessment of shoulder and arm symptoms before and after PEMF. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. Patients did not complete the necessary surveys assessing their shoulder and arm symptoms.
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Clinical Assessment of Shoulder and Arm Symptoms Before and After PEMF
Description: No participants were assessed for this secondary outcome measure: clinical assessment of shoulder and arm symptoms before and after PEMF. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. There was a lack of post-clinical assessment data as well as poor patient compliance with the 14 day mark follow up. Therefore, no meaningful results could be derived since there was no quantifiable means to compare before and after PEMF data points.
Time Frame: Pre- and Post-Operative Period
Population: No participants were assessed for this secondary outcome measure: clinical assessment of shoulder and arm symptoms before and after PEMF. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables due to lack of post-clinical assessment data and poor patient compliance with the 14 day mark follow up.
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Lymphedema
Description: No participants were assessed for this secondary outcome measure: lymphedema. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. No meaningful quantifiable data could be obtained on degree of lymphedema, and thus effect of PEMF intervention could not be analyzed.
Time Frame: Pre- and Post-Operative Period
Population: No participants were assessed for this secondary outcome measure: lymphedema. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. No meaningful quantifiable data could be obtained on degree of lymphedema, and thus effect of PEMF intervention could not be analyzed.
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Narcotic Pain Medications
Description: No participants were assessed for this secondary outcome measure: narcotic pain medications. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. Patients were instructed to complete logs at home indicating narcotic pain medications, and patients did not submit necessary logs assessing need for pain medications and level of nausea and vomiting; therefore, no meaningful data could be analyzed.
Time Frame: Post-Operative Period
Population: No participants were assessed for this secondary outcome measure: narcotic pain medications. No data was collected/calculated, and hence the data cannot be summarized to include in the data tables. Patients were instructed to complete logs at home indicating narcotic pain medications, and patients did not submit necessary logs.
Arm/Group | Sham PEMF Device | PEMF Device
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time frame for adverse event reporting was the time during which the PEMF device was on the patient, maximum 2 weeks.
Arm/Group | Sham PEMF Device | PEMF Device
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No